CLINICAL TRIAL: NCT06044974
Title: Piano Level Laser Therapy Versus Epidermal Growth Factor in the Treatment of Myogenic Tempromandibular Disorder (Randomized Clinical Trial)
Brief Title: Nd-YAG Laser Versus Epidermal Growth Factor For Myogenic Tempromandibular Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Passant Osama Qataya, Assistant Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ndyag laser december 2022
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Joint Disorders
Keywords: TMD; Laser; EGF; saliva; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Epidermal Growth Factor

STUDY DESIGN:
Intervention Model Description: Two groups suffering from myogenic Tempromandibular disorders. Each group will receive either photobiomodulation using ND-YAG laser or injection of epidermal growth factor intramuscular.
Who Masked: Outcomes Assessor
Masking Description: Data assessors: oral medicine co-worker and biochemist specialist, and statistician will all be blinded to the treatment of each patient; a triple-blinded clinical trial. Patients and primary clinician will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (n=15): combined therapy sessions using 1064 nm Nd-YAG laser (once/week) (Active Comparator): Each treatment session will include: a first pass, which will be performed using "cold" Piano Level Laser Therapy "PLLT" settings for photo biomodulation - MSP pulse (100 µs), P = 2W, 10 Hz, with 1 minute treatment duration per spot. A second pass, higher "warm" PLLT settings that causes mild heating of the tissue, aimed at pain relief - MSP pulses 5 W, 60 Hz, where the handpiece will be held at each spot from 30 seconds to 1 minute, depending on patient heat tolerance
  . Both the masseter and temporalis muscles will be divided into 3 spots: insertion, body, and origin for the masseter muscle and anterior, middle, and posterior for temporalis muscle. A stamping technique will be carried out for both passes.
  Interventions: Device: Nd-YAG Fotona
- Group II (n=15): Epidermal Growth factor (EGF) injection (Active Comparator): Epidermal Growth factor (EGF) injection into masseter and temporalis muscles. Each muscle will be divided into 3 zones; origin, body and insertion for masseter muscle, anterior, middle, and posterior for temporalis muscle
  * For masseter muscle injection, 3-point injection technique will be followed: 1 injection point in each zone. For temporalis muscle injection, 3-point injection technique will be followed: 1 in each zone
  * Each point will receive 0.1 ml of EGF
  Interventions: Drug: Epidermal Growth Factor

INTERVENTIONS:
Device: Nd-YAG Fotona — four combined therapy sessions using 1064 nm Nd-YAG laser (once/week)
  Arms: Group I (n=15): combined therapy sessions using 1064 nm Nd-YAG laser (once/week)
Drug: Epidermal Growth Factor — Epidermal growth factor "EGF-genesis" by Dermaquel Paris n into masseter and temporalis muscles. Each muscle will be divided into 3 zones; origin, body and insertion for masseter muscle, anterior, middle, and posterior for temporalis muscle
  Arms: Group II (n=15): Epidermal Growth factor (EGF) injection

SUMMARY:
A clinical trial comparing the potential effect of 2 different modalities (Nd-YAG Laser Versus Epidermal growth factor injection) on pain reduction in patients suffering from myogenic tempromandibular disorder.

DETAILED DESCRIPTION:
Background: Tempromandibular disorders (TMDs) form a public health issue and are considered the second most common musculoskeletal problem (after chronic lower back pain) causing pain and disability. Myogenic TMD is one of the commonly prevalent TMDs with unclear pathophysiology. Central and peripheral sensitization are thought to play an evident role in development of myogenous TMD. Many treatment modalities have been proposed to eliminate pain, improve function and quality of life. Laser photobiomodulation has gained popularity in pain therapy and in treatment of chronic painful musculoskeletal disorders, among which are TMDs. Piano level laser therapy (PLLT) enables delivering different high intensities using large spot sizes and can be considered beneficial in the treatment of painful myogenic TMD.

Epidermal growth factor (EGF) has been found to repair muscle damage and increase muscle quality through direct promotion of proliferation and differentiation of muscle cells in addition to regulating the inflammatory response. EGF can be another minimally invasive treatment modality for chronic painful myogenic TMD. Glutamate and nerve growth factor (NGF) are considered neuropeptides associated with pain and hyperalgesia.

They have been related to painful TMD and have also been detected in saliva of patients suffering from chronically painful conditions including TMDs. Aim: The present study aims to evaluate and compare the effectiveness of Piano level laser therapy using 1064nm Nd-YAG laser and intramuscular EGF injection in pain alleviation, improvement of function and quality of life in patients suffering from myogenic temporomandibular disorder. The impact of these treatment modalities on levels of salivary glutamate and nerve growth factor pain mediators will also be investigated. Materials and Methods: A randomized clinical trial will be carried out on 30 patients suffering from chronic painful myogenic TMD based on diagnostic criteria for temporomandibular disorders (DC/TMD). Group I (n=15 patients) will be treated using 1064 nm Nd-YAG Laser: in 4 combined (cold=2W, warm=5W) laser therapy sessions (once/week) using stamping technique on masseter and temporalis muscles. Group II (n=15 patients) will be treated by intramuscular injection of EGF in masseter and temporalis muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, both males and females, 20 years and older will be included in this clinical trial.
2. Patients suffering from myogenic TMD (myogenic TMD/ Myofascial pain without referral/ Myofascial pain with referral) based on Diagnostic criteria for diagnosis of Tempromandibular joint disorders (DC/TMD) criteria (1)
3. Patients suffering of unilateral or bilateral chronic pain (> 3 months duration) related to masseter and temporalis muscles (29)
4. Patients that have not responded to conservative modes of treatment (analgesics, muscle relaxants, fomentation, splints ect.).

Exclusion Criteria:

* Patients suffering from any condition that could alter pain sensitivity; neurological diseases, pain of dental origin, pregnancy or lactation, high blood pressure, diabetes mellitus, rheumatic inflammatory disease, fibromyalgia, obstructive sleep apnea, skin infection over injection areas related to masseter and temporalis muscles, and restrictions for the use of laser (pacemakers) (6, 20, 30) 2. Participants on medications that can affect pain sensitivity and pain perception; anticoagulants, analgesics, antidepressants during the last 2 weeks before the study (6, 20) 3. Smokers or those with conditions that could affect saliva collection or composition; hyposalivation, poor oral hygiene, periodontitis and oral mucosal diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Pain Score (Numerical Rating Scale) | Pain will be measured at baseline, 7,14,21 days, and 4, 12 weeks.
  Subjective Pain score as measured by Numerical Rating Scale (NRS) on a scale from "0" to "10", where "0" means no pain at all and "10" means worst response and maximum pain.

SECONDARY OUTCOMES:
Quality of Life using Oral Health Impact Profile (OHIP)-14 questionnaire | baseline, and 4, 12 weeks
  Quality of life questionnaire using OHIP-14 questionnaire, a score from 0 to 14, where score "0" means best quality of life impact and score "14" means the worst impact on quality of life.
Maximum unassisted opening | baseline, 7, 14, 21 days, and 4, 12 weeks.
  Maximum unassisted opening even if associated with pain measured in mm or cm
Pain Free Opening | baseline, 7, 14, 21 days, and 4, 12 weeks.
  Pain free opening measured in mm or cm
Salivary levels of glutamate | baseline, and 4, 12 weeks
  Detection of salivary pain mediators using enzyme-linked immunosorbent assay (ELISA) technique
Salivary levels of Nerve growth factor | baseline, and 4, 12 weeks
  Detection of salivary pain mediators using enzyme-linked immunosorbent assay (ELISA) technique

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: October 2023
Access Criteria: clinicaltrials.gov
URL: http://clinicaltrials.gov

REFERENCES:
- [Derived] Qataya PO, Zaki AM, Amin F, Swedan A, Elkafrawy H. Effect of Nd-YAG Laser Versus Epidermal Growth Factor Injection on Salivary Pain Mediators in Myogenic Temporomandibular Disorders (A Randomized Clinical Trial). J Oral Pathol Med. 2025 Nov;54(10):992-1000. doi: 10.1111/jop.70053. Epub 2025 Sep 2. PMID 40891771